CLINICAL TRIAL: NCT03103763
Title: ATIVO Study - Anticoagulation Therapy in the Very Old
Brief Title: Anticoagulation Therapy in the Very Old
Acronym: ATIVO
Status: Completed | Type: Observational
Sponsor: Robert Stein (Other)
Responsible Party: Sponsor-Investigator, Robert Stein, Medical Director of Anticoagulation Services, MaineHealth
Organization: MaineHealth (Other)
Other Study IDs: PenobscotBMC
Record Dates: First submitted 2017-04-01; First posted 2017-04-06 (Actual); Results first posted 2020-06-16 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Atrial Fibrillation
Keywords: Elderly; Anticoagulation; Risk Assessment
MeSH Terms: conditions — Atrial Fibrillation | interventions — Warfarin; Vitamin B 6

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Aged 90 and older: Subjects 90 years and older with atrial fibrillation, taking warfarin, followed by the Penobscot Bay Medical Center Anticoagulation Services.
  Interventions: Drug: Warfarin
- Aged 80-89: Subjects aged 80-89 with atrial fibrillation, taking warfarin, followed by the Penobscot Bay Medical Center Anticoagulation Services.
  Interventions: Drug: Warfarin
- Aged 70-79: Subjects aged 70-79 with atrial fibrillation, taking warfarin, followed by the Penobscot Bay Medical Center Anticoagulation Services.
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Warfarin — Patients on warfarin for atrial fibrillation
  Other Names: Coumadin, Jantoven

SUMMARY:
This study is designed to evaluate the efficacy and safety of warfarin anticoagulation in the very old and attempt to identify risk factors which may impede safe and effective anticoagulation.

DETAILED DESCRIPTION:
This is a prospective registry study with data being collected continuously for 24 months.

Patients who have electrocardiographically confirmed atrial fibrillation, are being followed by the Pen Bay Medical Center Anticoagulation Services and are at least 90 years old will be recruited into the study. A matched cohort of patients between the ages of 80 and 89 and another matched cohort of patients between the ages of 70 and 79 will also be recruited into the study for comparison.

Data related to adverse events, concomitant medications, living arrangements, mobility and alcohol use will be collected every 6 months. In addition the CHA2DS2-VASc (score for atrial fibrillation stroke risk), HAS - BLED (major bleeding risk score for patients on anticoagulation), frailty and Mini Cog scores will be recalculated at each visit.

ELIGIBILITY:
Inclusion Criteria:

* 70 years of age or older
* electrocardiographically confirmed atrial fibrillation
* anticipated regular follow up with patient by Penobscot Bay Medical Center (PBMC) Anticoagulation Services
* Subject or legally authorized representative must be willing to provide informed consent

Exclusion Criteria:

- Patients not being followed by the PBMC Anticoagulation Services

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All patients seen by the PBMC Anticoagulation Services who are taking warfarin, have atrial fibrillation aged 90 years and older will be invited to participate in the study. A matched cohort of patients aged 80-89 will also be enrolled as well as another matched cohort of patients aged 70-79 who are on warfarin for atrial fibrillation will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2019-09-03 (Actual); Study Completion 2019-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert W. Stein, MD, Principal Investigator — MaineHealth
Locations (1):
- Penobscot Bay Medical Center, Rockport, Maine, United States

IPD SHARING:
Plan to Share IPD: No
date will not be shared

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aged 90 and Older | Aged 80-89 | Aged 70-79
Started | 44 | 44 | 44
Completed | 29 | 36 | 37
Not Completed | 15 | 8 | 7
Not completed — Death | 15 | 5 | 5
Not completed — Withdrawal by Subject | 0 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aged 90 and Older | Aged 80-89 | Aged 70-79 | Total
Number analyzed (Participants) | 44 | 44 | 44 | 132
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 44 | 44 | 44 | 132
Age, Continuous [Mean (Full Range); unit: years] | 93 [90 to 100] | 84 [80 to 89] | 74 [70 to 79] | 84 [70 to 100]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 25 | 23 | 79
  Male | 13 | 19 | 21 | 53
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 44 | 44 | 44 | 132
Region of Enrollment [Number; unit: participants]
  United States | 44 | 44 | 44 | 132
Living at home alone [Count of Participants; unit: Participants] | 11 | 18 | 9 | 38
Living at home with paid help [Count of Participants; unit: Participants] | 2 | 2 | 1 | 5
Living at home with family [Count of Participants; unit: Participants] | 27 | 24 | 34 | 85
Living in assisted living [Count of Participants; unit: Participants] | 4 | 0 | 0 | 4
Living in Long Term Care [Count of Participants; unit: Participants] | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Experiencing Stroke
Description: Every 6 months the medical record was reviewed for evidence of stroke of any cause.
Time Frame: 24 months
Population: Three subjects in the 80-89 age group and two subjects in the 70-79 age group withdrew consent prior to end of study.
Measure: Count of Participants; unit: Participants
Arm/Group | Aged 90 and Older | Aged 80-89 | Aged 70-79
Number analyzed (Participants) | 44 | 41 | 42
Participants | 2 | 2 | 0

2. Primary Outcome: Number of Patients Experiencing a Major Bleeding Event
Description: defined as one of the following: fatal bleeding, symptomatic bleeding in a critical area or organ or bleeding causing a fall in hemoglobin of 2 g/dl or more or leading to a transfusion of 2 or more units of whole blood or red cells
Time Frame: 24 months
Population: Three subjects in the 80-89 age group and two subjects in the 70-79 age group withdrew consent prior to end of study.
Measure: Count of Participants; unit: Participants
Arm/Group | Aged 90 and Older | Aged 80-89 | Aged 70-79
Number analyzed (Participants) | 44 | 41 | 42
Participants | 4 | 2 | 4

3. Secondary Outcome: Number of Patients Experiencing a Traumatic Subdural Hemorrhage
Description: Number of subjects who experienced a traumatic subdural hemorrhage in each age group
Time Frame: 24 months
Population: Three subjects in the 80-89 age group and two subjects in the 70-79 age group withdrew consent prior to end of study.
Measure: Count of Participants; unit: Participants
Arm/Group | Aged 90 and Older | Aged 80-89 | Aged 70-79
Number analyzed (Participants) | 44 | 41 | 42
Participants | 0 | 0 | 0

4. Secondary Outcome: Number of Patients Experiencing a Traumatic Intracerebral Hemorrhage
Description: Number of subjects who experienced a traumatic intracerebral hemorrhage in each age group
Time Frame: 24 months
Population: Three subjects in the 80-89 age group and two subjects in the 70-79 age group withdrew consent prior to end of study.
Measure: Count of Participants; unit: Participants
Arm/Group | Aged 90 and Older | Aged 80-89 | Aged 70-79
Number analyzed (Participants) | 44 | 41 | 42
Participants | 0 | 0 | 0

5. Secondary Outcome: Number of Hospitalizations Patients Experienced
Description: Every 6 months the medical record was reviewed for any hospitalizations experienced by the subject within our healthcare system.
Time Frame: 24 months
Population: Three subjects in the 80-89 age group and two subjects in the 70-79 age group withdrew consent prior to end of study.
Measure: Number; unit: hospitalizations
Arm/Group | Aged 90 and Older | Aged 80-89 | Aged 70-79
Number analyzed (Participants) | 44 | 41 | 42
hospitalizations | 51 | 41 | 41

6. Secondary Outcome: Number of Patients Experiencing Cardiovascular Death
Description: Every 6 months the medical record was reviewed. All deaths were researched for cause and noted if the cause was related to the cardiovascular system.
Time Frame: 24 months
Population: Three subjects in the 80-89 age group and two subjects in the 70-79 age group withdrew consent prior to end of study.
Measure: Count of Participants; unit: Participants
Arm/Group | Aged 90 and Older | Aged 80-89 | Aged 70-79
Number analyzed (Participants) | 44 | 41 | 42
Participants | 15 | 5 | 5

7. Secondary Outcome: Number of Patients Experiencing Death Related to Anticoagulation
Description: All deaths were reviewed in the medical record to determine the cause and if it was related in any way to the use of anticoagulation therapy.
Time Frame: 24 months
Population: Three subjects in the 80-89 age group and two subjects in the 70-79 age group withdrew consent prior to end of study.
Measure: Count of Participants; unit: Participants
Arm/Group | Aged 90 and Older | Aged 80-89 | Aged 70-79
Number analyzed (Participants) | 44 | 41 | 42
Participants | 0 | 0 | 0

8. Secondary Outcome: Mean Time in Therapeutic Range at End of Study Participation
Description: International Normalized Ratio (INR) time in therapeutic range at the end of the individual's study participation.
Time Frame: up to 24 months
Population: All subjects were included in this analysis.
Measure: Mean (Standard Deviation); unit: percent of time in therapeutic range
Arm/Group | Aged 90 and Older | Aged 80-89 | Aged 70-79
Number analyzed (Participants) | 44 | 44 | 44
percent of time in therapeutic range | 72 (17) | 76 (18) | 70 (17)

ADVERSE EVENTS:
Time Frame: Because the study is a registry, no events were collected as adverse events. Outcomes were collected. All cause mortality was collected from date of consent up to 24 months.
Description: Death information was available. However, serious and other adverse event data were not monitored.
Arm/Group | Aged 90 and Older | Aged 80-89 | Aged 70-79
All-Cause Mortality (participants affected / at risk) | 15/44 | 5/41 | 5/42
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The small sample size limits the power of this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2018-12-13): https://cdn.clinicaltrials.gov/large-docs/63/NCT03103763/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-13): https://cdn.clinicaltrials.gov/large-docs/63/NCT03103763/SAP_001.pdf
  • Informed Consent Form (2017-03-20): https://cdn.clinicaltrials.gov/large-docs/63/NCT03103763/ICF_002.pdf